CLINICAL TRIAL: NCT03962075
Title: Short-term Outcomes of Laparoscopic Repair of Paravaginal Defects: A Clinical Trial
Brief Title: Short-term Outcomes of Laparoscopic Repair of Paravaginal Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hossam mohamed, principal investigator, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2765/20-6-2016
Record Dates: First submitted 2019-05-07; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Prolapse, Vaginal; Paravaginal Cystocele
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laparoscopic paravaginal repair (Other): patient enrolled in this arm were offered laparoscopic paravaginal repair by Using a 10mm laparoscope, video camera, was introduced through the umbilical trocar. Another 5 mm in suprapubic area and two 10 mm trocars in right and left lateral abdominal sides were introduced. The larger trocar was needed to accommodate the passage of needles into the abdomen. Spacing of trocars sufficiently from each other was needed to facilitate laparoscopic suturing. Transperitoneal approach to retropubic space was used. Two to four polypropylene sutures were applied on each side. Sutures were tied with intracorporeal technique All cases received diclofenac potassium 100 mg and meperidine hydrochloride 50 mg intramuscular with anesthesia recovery and 12 hours later second dose of diclofenac potassium was given. Also 40-60 mg Enoxaparin was given 6-12 hours postoperatively as subcutaneous injection.
  Foley's catheter was removed 6 hours postoperative
  Interventions: Procedure: laparoscopic paravaginal repair

INTERVENTIONS:
Procedure: laparoscopic paravaginal repair — Using a 10mm laparoscope, with video camera, was introduced through the umbilical trocar. Another 5 mm in suprapubic area and two 10 mm trocars in right and left lateral abdominal sides were introduced. The larger trocar was needed to accommodate the passage of needles into the abdomen. Spacing of trocars sufficiently from each other was needed to facilitate laparoscopic suturing. Transperitoneal approach to retropubic space was used. Two to four polypropylene sutures were applied on each side. Sutures were tied with intracorporeal technique

SUMMARY:
this study designed To evaluate the efficacy and outcomes of laparoscopic approach for repair of paravaginal defects associated with anterior vaginal wall prolapse.

DETAILED DESCRIPTION:
This prospective interventional study. designed to evaluate the efficacy and outcomes of laparoscopic approach for repair of paravaginal defects associated with anterior vaginal wall prolapse .fifty participants with cystocele of lateral type offered laparoscopic paravaginal repair. the investigator used a 10mm laparoscope, with video camera, was introduced through the umbilical trocar. Another 5 mm in suprapubic area and two 10 mm trocars in right and left lateral abdominal sides were introduced. The larger trocar was needed to accommodate the passage of needles into the abdomen. Spacing of trocars sufficiently from each other was needed to facilitate laparoscopic suturing. Transperitoneal approach to retropubic space was used. Two to four polypropylene sutures were applied on each side. Sutures were tied with intracorporeal . The study evaluated the following outcomes Operative time, intra-operative blood loss, hospital stay , post-operative urinary symptoms, post-operative pain, fever, haematuria, post-operative vaginal wall prolapse .

ELIGIBILITY:
Inclusion Criteria:

* female patient with cystocele of lateral type ( paravaginal defect )

Exclusion Criteria:

* previous retropubic surgery,
* uterine prolapse,
* stress urinary incontinence or
* morbid obesity

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patient complaining of anterior vaginal wall prolapse of lateral type
Enrollment: 50 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
operative time | insertion of the primary tracer ( umbilical trocar )-during the procedure - ends with removing camera telescope
  time needed for the procedure to be completed
intraoperative blood loss | start with dissection or retropubic space - during the procedure -ends with removing the camera telescope at the end of operation
  amount of bleeding during the procedure
post-operative pain: Faces Pain Scale | start after patient recovery from anaesthesia - ends after 12 hours
  assessment of pain using Faces Pain Scale( displaying faces that show how much pain the participant can feel. starting with the face on far left shows no pain as The faces move to the right show more and more pain that ends with the face on the right which shows the worst pain then the participants Point to the face that shows how much they feel pain , Each face has a score 0, 2, 4, 6, 8, or 10, so score "0" = "no pain" and score "10" = "very much pain).
post-operative hematuria | starts observation of urine 1hour after end of operation - ends 24 hours after the starting observation
  visible red or brown discoloration of urine .
hospital stay | during hospitalization
  hours needed to keep the patient in hospital post operative
fever | starts after shifting the patient from the recovery room to inpatient ward - end 24 hours after shifting the patient
  body temperature 38 Celsius or above

SECONDARY OUTCOMES:
post-operative vaginal wall prolapse | starts one week following the procedure - three months after the procedure - six months after the procedure -ends one year after the procedure
  assessment of the anterior vaginal wall using:Pelvic Organ Prolapse Quantification System .
post-operative abnormal urinary symptoms | starts one week following the procedure - three months after the procedure - six months after the procedure -ends one year after the procedure
  abnormal urinary symptoms: ( inability to urinate voluntary- pain during micturition - involuntary escape of urine )